CLINICAL TRIAL: NCT01095653
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin as Monotherapy in Asian Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet and Exercise
Brief Title: A Phase III Study of BMS-512148 (Dapagliflozin) in Asian Patients With Type 2 Diabetes Who Are Not Well Controlled With Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: AstraZeneca, Bristol-Myers Squibb (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB102-054
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Metformin; Drug: Dapagliflozin Placebo
- Group 2 (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Metformin; Drug: Dapagliflozin Placebo
- Group 3 (Experimental)
  Interventions: Drug: Metformin; Drug: Dapagliflozin Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 5 mg, Once daily, 24 weeks
  Other Names: BMS-512148
  Arms: Group 1
Drug: Dapagliflozin — Tablets, Oral, 10 mg, Once daily, 24 weeks
  Other Names: BMS-512148
  Arms: Group 2
Drug: Metformin — Tablets, Oral, 500-2000 mg (as needed for rescue based on protocol specific criteria), Up to 20 weeks
  Other Names: Glucophage®
Drug: Dapagliflozin Placebo — Tablets, Oral, 0 mg, Once daily, 24 weeks

SUMMARY:
The purpose of this clinical research study is to learn if BMS-512148 (Dapagliflozin) can improve (decrease) blood glucose values in Asian patients with Type 2 Diabetes who have never been treated with medication or have been on medication for less than 24 weeks since their original diagnosis of Diabetes. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years old, with type 2 diabetes and with inadequate glycemic control
* Drug naive or treated with anti-diabetic medication for < 24 weeks
* C-peptide ≥ 1.0 ng/mL
* Body Mass Index ≤ 45.0 kg/m²

Exclusion Criteria:

* AST and/or ALT > 3 times ULN
* Serum total bilirubin > 2 mg/dL
* Serum creatinine ≥ 1.50 mg/dL for men or ≥ 1.40 mg/dL for women
* Creatine kinase ≥ 3 times ULN
* Symptoms of severely uncontrolled diabetes
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncological, endocrine, psychiatric, or rheumatic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1179 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (28):
- China (17):
  - Local Institution, Hefei, Anhui
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Guanzhou, Guangdong
  - Local Institution, Wuhan, Hubei
  - Local Institution, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Wuxi, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Beijing
  - Local Institution, Wuhan
  - Local Institution, Xi'an
- India (4):
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Indore, Madhya Pradesh
  - Local Institution, Bangalore
  - Local Institution, Jaipur
- South Korea (4):
  - Local Institution, Seoul, Nowon-GU
  - Local Institution, Busanjin-gu
  - Local Institution, Guri-si
  - Local Institution, Seoul
- Taiwan (3):
  - Local Institution, Taichung
  - Local Institution, Taipei
  - Local Institution, Yung Kang City

REFERENCES:
- See also: Publication — https://www.ncbi.nlm.nih.gov/pubmed?term=%22Clinical+therapeutics%22%5BJour%5D+AND+2014%5Bpdat%5D+AND+Dapagliflozin&TransSchema=title&cmd=detailssearch&_sm_au_=iFHnRDqNTf1p01TQ

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 1179 participants enrolled, 514 completed a qualification period. Of these 514 participants, 393 were randomized and received treatment. Of these 393 participants, 343 completed double-blind treatment period.
Groups:
- Placebo: Participants received dapagliflozin matching placebo once daily for up to 24 weeks (may include the addition of open-label metformin as rescue)
- Dapagliflozin 5 mg: Participants received dapagliflozin 5 mg once daily for up to 24 weeks (may include the addition of open-label metformin as rescue)
- Dapagliflozin 10 mg: Participants received dapagliflozin 10 mg once daily for up to 24 weeks (may include the addition of open-label metformin as rescue)
Period: Overall Study
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Started | 132 | 128 | 133
Completed | 113 | 113 | 117
Not Completed | 19 | 15 | 16
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 4
Not completed — Lost to Follow-up | 1 | 0 | 4
Not completed — Withdrawal by Subject | 4 | 5 | 3
Not completed — non-compliance, not met criteria, etc. | 10 | 6 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg | Total
Number analyzed (Participants) | 132 | 128 | 133 | 393
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (10.87) [20 to 75] | 53.0 (11.07) [29 to 79] | 51.2 (9.89) [21 to 72] | 51.3 (10.67) [20 to 79]
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 120 | 108 | 123 | 351
  65 to younger than 75 years | 11 | 14 | 10 | 35
  75 years and older | 1 | 6 | 0 | 7
Sex/Gender, Customized [Number; unit: Participants]
  Male | 87 | 84 | 86 | 257
  Female | 45 | 44 | 47 | 136
Race/Ethnicity, Customized [Number; unit: Participants]
  ASIAN INDIAN | 8 | 8 | 9 | 25
  CHINESE | 117 | 114 | 117 | 348
  JAPANESE | 1 | 0 | 1 | 2
  KOREAN | 5 | 6 | 5 | 16
  ASIAN OTHER | 1 | 0 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 72.18 (13.234) | 68.89 (11.429) | 70.92 (11.637) | 70.68 (12.177)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.93 (3.644) | 25.17 (3.285) | 25.76 (3.434) | 25.62 (3.465)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 24 (Last Observation Carried Forward [LOCF])
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 4, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing HbA1c values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: % of hemoglobin
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 127 | 122 | 127
% of hemoglobin | -0.29 (0.0681) | -1.04 (0.0695) | -1.11 (0.0680)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Primary endpoints were tested at alpha=0.027 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-0.94 to -0.56], Standard Error of Mean 0.0975
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Primary endpoints were tested at alpha=0.027 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.01 to -0.63], Standard Error of Mean 0.0962

2. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Fasting plasma glucose was measured as milligrams per deciliter(mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing FPG values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 131 | 127 | 128
mg/dL | 2.5 (2.237) | -25.1 (2.274) | -31.6 (2.255)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -27.7, 95% CI 2-sided [-34.0 to -21.4], Standard Error of Mean 3.203
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -34.2, 95% CI 2-sided [-40.4 to -27.9], Standard Error of Mean 3.174

3. Secondary Outcome: Adjusted Mean Change From Baseline in 2-hour Post Liquid Meal Glucose (PLMG) (mg/dL) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Post Liquid Meal Glucose was measured as milligrams per deciliter(mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. PLMG measurements were obtained on Day 1 and week 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing PLMG values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 105 | 100 | 105
mg/dL | 1.08 (4.5663) | -46.8 (4.6559) | -54.9 (4.5257)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -47.9, 95% CI 2-sided [-60.80 to -34.96], Standard Error of Mean 6.5667
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -56.0, 95% CI 2-sided [-68.66 to -43.28], Standard Error of Mean 6.4489

4. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight (kg) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 8, 12, 16, 20, and 24 of the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing body weight values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 132 | 128 | 128
kg | -0.27 (0.2279) | -1.64 (0.2315) | -2.25 (0.2308)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-2.01 to -0.73], Standard Error of Mean 0.3259
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.62 to -1.34], Standard Error of Mean 0.3242

5. Secondary Outcome: Percentage of Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <7.0% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Percent adjusted for baseline HbA1c. Therapeutic glycemic response is defined as HbA1c <7.0%. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin. Mean and standard error for percentage of participants were estimated by modified logistic regression model.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: Percentage of participants
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 127 | 122 | 127
Percentage of participants | 21.3 (3.310) | 42.6 (4.300) | 49.8 (4.032)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, Modified logistic regression — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = 21.3, 95% CI 2-sided [11.1 to 31.6], Standard Error of Mean 5.238
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; p < 0.0001, Modified logistic regression — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = 28.5, 95% CI 2-sided [18.6 to 38.3], Standard Error of Mean 5.022

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of double-blind treatment 24 weeks plus 4 days for non-serious adverse event; plus 30 days for serious adverse event.
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Serious Adverse Events (participants affected / at risk) | 2/132 | 5/128 | 4/133
Other Adverse Events (participants affected / at risk) | 38/132 | 28/128 | 23/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=132) | Dapagliflozin 5 mg (N=128) | Dapagliflozin 10 mg (N=133)
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
GOITRE (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
URETHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=132) | Dapagliflozin 5 mg (N=128) | Dapagliflozin 10 mg (N=133)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 14 (14) | 10 (10) | 9 (9)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 (13) | 10 (10) | 9 (13)
NASOPHARYNGITIS (Infections and infestations) | 5 (5) | 7 (8) | 4 (6)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 7 (7) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No